CLINICAL TRIAL: NCT02389595
Title: Selection of a Protective T Cell-based HIV-1/FIV Vaccine Devoid of Viral Enhancing Epitopes
Brief Title: Selection of a Protective T Cell-based HIV-1/FIV Vaccine
Status: Active, not recruiting | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201401012-N
Record Dates: First submitted 2015-03-10; First posted 2015-03-17 (Estimated); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: HIV
Keywords: HIV; vaccine; T cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum Whole Blood T cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HIV positive subjects: This group will provide a blood sample.
  Interventions: Other: HIV positive subjects
- Non-infected control subjects: This group consist of de-identified blood samples from a commercial source.
  Interventions: Other: Non-infected control subjects

INTERVENTIONS:
Other: HIV positive subjects — This group will provide a blood sample.
  Groups: HIV positive subjects
Other: Non-infected control subjects — This group will be de-identified blood samples from a commercial source.
  Groups: Non-infected control subjects

SUMMARY:
The purpose of this research study is to develop a vaccine against Human immunodeficiency virus (HIV), a disease that causes AIDS in people,. The investigator will be looking at viruses similar to HIV in animals. Since these viruses are very similar to HIV, the blood from humans who have been exposed to HIV will be tested to see if the immune system will recognize the HIV and prevent infection.

HIV targets the immune system by attacking certain T cells called CD4+ T cells. There are parts on the AIDS viruses that help the virus infect these cells and other parts that help the immune system prevent viral infection by activating protective T-cells that fight HIV. Different T-cell populations are very important in most vaccines as they act as "effectors" that work as part of the immune system to recognize and fight off HIV infection. When effector T cells are activated by appropriate "protective" part(s) of the virus they either block HIV from reproducing or kill HIV infected cells. By finding these common protective parts of each of these human and animal AIDS viruses, the investigator hopes to make a vaccine that helps the immune system prevent HIV infection by avoiding parts that attack CD4+ T cells and may worsen HIV infection and selecting for parts that stimulate effector T cells that fight HIV infection.

DETAILED DESCRIPTION:
As a participant in this study a blood drawn will performed.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between 18 and 65 years old who are HIV positive

Exclusion Criteria:

* Persons with other immune diseases that would result in autoimmunity or aberrant immune responses (such as subjects who have undergone chemotherapy within the past year).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV positive individuals between 18 and 65 years old
Sampling Method: Non-Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2015-05 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
T cell proliferation in response to viral epitopes | 120 hours (5 days)

SECONDARY OUTCOMES:
Cytokine production in response to viral epitopes | 24 hours (1 day)
Cytotoxin production in response to viral epitopes | 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Janet K Yamamoto, PhD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - University of Florida, Gainesville, Florida
  - UF Center for AIDS Research Education and Service, Jacksonville, Florida